CLINICAL TRIAL: NCT05159830
Title: Cannabidiol for Reducing Drinking in Alcohol Use Disorder and Modifying the Effects of Alcohol on the Brain and the Liver: a Phase 2 Clinical Trial.-The CARAMEL Study
Brief Title: Cannabidiol for Reducing Drinking in Alcohol Use Disorder
Acronym: CARAMEL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-004740-30
Record Dates: First submitted 2021-09-20; First posted 2021-12-16 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: CARAMEL is a phase-2, national, multi-site, interventional (category 1), double-blind, randomized, placebo-controlled trial, conducted in 76 subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: CLEAVER LEAVES - ECOMEDICS SAS produce Oral oil of Cannabidiol and Placebo of similar galenic form. They will be responsible for the pharmaceutical analyses of the product.
  Eurofins-LC2 will import the oral oil after authorization from the ANSM, and will relabeled individual vials for each participant, and regular dispatching into the hospital pharmacy.
  Local hospital pharmacies will be in charge to deliver treatment individual vials to the investigators for dispensing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): CBD Group from 20mg x 2/day up to 600mg/day
  Interventions: Drug: Cannabidiol oral oil
- PLACEBO (PCB) (Placebo Comparator): PCB Group from 20mg x 2/day up to 600mg/day
  Interventions: Drug: Placebo oral oil

INTERVENTIONS:
Drug: Cannabidiol oral oil — The CBD dosing used in the CARAMEL study will start at 40mg/d up to 600 mg/d. Oral oil contain 20 mg of CBD. 20 mg because our supplier does not have a more highly dosed oral oil.
  Arms: Cannabidiol (CBD)
Drug: Placebo oral oil — Placebo of similar cannabidiol galenic form
  Arms: PLACEBO (PCB)

SUMMARY:
The non-psychotomimetic cannabis compound cannabidiol (CBD) has been found effective for reducing alcohol drinking in mice. Moreover, other experimental studies have found that CBD reduced alcohol-induced steatosis in the liver, and reduced alcohol-related injury in the brain. Despite these promising results from animal data, no human study has been conducted yet in alcohol use disorder (AUD).

DETAILED DESCRIPTION:
CBD has several potential therapeutic prospects in AUD. Preclinical studies now support the potential of CBD for drinking reduction in AUD subjects. Moreover, other experimental studies have found that CBD reverse the alcohol-induced steatosis process in the liver. These two experimental effects need a translational confirmation in humans through an explanatory phase 2 study. In addition, CBD could also exert neuroprotective effects that reduce the deleterious effects of alcohol on the brain. In both the liver and the brain, the idiosyncratic anti-inflammatory effects of CBD could thus strengthen the overall harm reduction allowed by drinking reduction in AUD ± ALD patients.

CBD deserves an exploratory study assessing whether the different therapeutic prospects in AUD are warranted. Moreover, because CBD is extracted from cannabis, and even if it is a CB1 antagonist with no psychotomimetic effects and no reported potential for abuse, the first pieces of evidence in AUD should confirm that CBD is safe in AUD subjects.

The CARAMEL study is a phase-2 clinical trial on 76 subjects, which aims to investigate the efficacy of CBD on reducing alcohol drinking, as well as the potential of CBD for restraining alcohol-induced brain and liver injuries, and confirm the good safety profile of CBD.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18 - 65 years
* Being fluent in French
* Having read the information procedure and signed the informed consent sheet.
* Being affiliated with health insurance.
* DSM-5 criteria for AUD (all stages) (American Psychiatric Association, 2013)
* Average drinking level of at least 12 standard-drinks (120g of ethanol) per day over the month prior to inclusion (i.e., a total alcohol consumption of 336 standard-drinks during the 28-day assessment period prior to inclusion), using the A-TLFB.

Exclusion Criteria:

* At least one day of abstinence (no alcohol drinking) during the month prior to inclusion
* Criteria for liver cirrhosis (Child-Pugh B or C)
* DSM-5 criteria for schizophrenia, schizoaffective disorder, or bipolar disorder, using the MINI 7.0.2.
* Current suicidality, using the MNI 7.0.2
* Lifelong history of suicide attempts
* Lifelong history or current DSM-5 criteria for substance use disorder (other than alcohol or nicotine) using the MINI 7.0.2.
* Any detected use of cannabis or any other cannabinoid within 60 days prior to screen
* Patients with transaminase elevations greater than 3 times upper the limit of normal and bilirubin greater than 2 times upper the limit of normal.
* Impaired medical condition (investigator's decision)
* Pregnancy, lactation, or insufficient contraceptive measure (precautionary measure) (See 5.2 for acceptable birth control methods)
* Patients with cancer, HIV, pulmonary arterial hypertension, epilepsy and with rifampicin, St. John's wort, Mammalian target of rapamycin (mTOR), calcineurin inhibitors or triazole antifungal agents like posaconazole, fluconazole… .
* History of vascular accident and/or cardiac arrhythmias and/or myocardial infarction
* Patients receiving acamprosate, naltrexone, disulfiram, nalmefene, topiramate, baclofen for AUD within 30 days prior to screening.
* MRI contraindication: pacemaker, insulin pump, heart metal valve, cochlear implant…
* Known hypersensitivity to the active principle (cannabidiol) or excipients (sucralose, menthol, mannitol).
* Person under tutorship or curatorship.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the total consumption of alcohol (in standard-drinks, sd) in the 28 last days (week 8 to week 12) of the study, using the Alcohol Timeline Followback (A-TLFB) daily self-report of alcohol drinking | Five months
  The difference between the total alcohol consumption during 28 days preceding the study, and the 28 last days of the study, will be compared between the two groups.

SECONDARY OUTCOMES:
Difference (i.e., inclusion minus end of study) in alcohol craving scores using the Obsessive Compulsive Drinking Scale (OCDS). | Five months
  Inclusion minus end of study using the OCDS. The Obsessive Compulsive Drinking Scale (OCDS) is a 14-item questionnaire that measures an individual's alcohol use and his/her attempts to control his/her drinking. Each item is scored on a scale from 0 to 4.Obsessive subscale is the summation of items 1-6.Compulsive subscale is the summation of items 7-14.
Difference in alcohol use disorder scores using the Alcohol Use Disorders Identification Test scale (AUDIT-C). | Five months
  inclusion minus end of study The Alcohol Use Disorders Identification Test (AUDIT-C) is an alcohol screen that can help identify patients who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence).
  Probable misuse: score > 4 for men and > 3 for women. Probable dependence: score > 10 regardless of sex.
Difference in anxiety and depression Hospital Anxiety and Depression Scale (HADS) | Five months
  Inclusion minus end of study Each answer corresponds to a number. By adding these numbers, we obtain a total score per column (anxiety and depression). If the score of a column is greater than or equal to 11, it means that the subject suffers from anxiety or depression
Difference in Controlled Attenuation Parameter (CAP) scores | Five months
  Inclusion minus end of study Using ultra-sound electrography which measures liver steatosis using transient ultra-sound elastography, between V0 and V4
Change in steatosis scores between V0 and V4, using Proton Density Fat Fraction (PDFF) estimated on the structural liver based on Chemical Shift Encoding-MRI (CSE-MRI) and MR Spectroscopy (MRS). | Five months
  Inclusion minus end of study
Between-group comparison of recovery of grey matter integrity in corticostriatal-limbic circuits, between V0 and V4, using MRI Voxel Based Morphometry (VBM) and cortical thickness measures. | Five months
  Inclusion minus end of study

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin ROLLAND, MD, PhD, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No